CLINICAL TRIAL: NCT02398188
Title: A Multi-Center, Randomized, Double-Blinded, Placebo-Controlled Study Evaluating the Safety and Efficacy of LIPO-202 for the Reduction of Central Abdominal Bulging Due to Subcutaneous Fat in Non-Obese Subjects
Brief Title: Evaluating the Safety and Efficacy of LIPO-202 for the Reduction of Central Abdominal Bulging Due to Subcutaneous Fat (AbCONTOUR2)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Evofem Inc. (Industry)
Collaborators: Neothetics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LIPO-202-CL-19
Record Dates: First submitted 2015-03-19; First posted 2015-03-25 (Estimated); Results first posted 2019-01-07 (Actual); Last update posted 2019-01-07 (Actual); Status verified 2018-10

CONDITIONS: Central Abdominal Bulging
MeSH Terms: interventions — Salmeterol Xinafoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- LIPO-202 (Experimental): Experimental arm
  Interventions: Drug: LIPO-202
- Placebo (Placebo Comparator): Placebo comparator
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LIPO-202
  Other Names: Salmeterol
  Arms: LIPO-202
Drug: Placebo
  Other Names: Placebo for LIPO-202
  Arms: Placebo

SUMMARY:
This is a multi-center, randomized, double-blinded, placebo-controlled study evaluating the safety and efficacy of LIPO-202 for the reduction of central abdominal bulging due to subcutaneous fat in non-obese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or non-pregnant female subjects
* Capable of providing written consent.
* BMI < 30 kg/m2
* Stable diet and exercise routine
* Central abdominal bulging that is evaluated by the clinician at least slight bulge, not flat

Exclusion Criteria:

* Have had any treatment of the fat around your abdomen, including surgical procedures (tummy tuck, liposuction), injections for fat loss or treatments with devices to reduce fat in your abdomen.
* Plan on starting a weight loss or exercise program during the study.
* Known hypersensitivity to study drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 793 (Actual)
Dates: Start 2015-04-09 (Actual); Primary Completion 2015-10-29 (Actual); Study Completion 2015-10-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Feldman, Study Director — Neothetics, Inc
Locations (35):
- United States (35):
  - Total Skin and Beauty Dermatology Center, Birmingham, Alabama
  - Stoll Dermatology of Beverly Hills, Beverly Hills, California
  - Diagnamics, Inc., Encinitas, California
  - Ablon Skin Institute And Research Center, Manhattan Beach, California
  - Dermatology Specialists, Inc., Oceanside, California
  - Rancho Mirage Dermatology, Rancho Mirage, California
  - Faces Plus, San Diego, California
  - Therapeutics Clinical Research, San Diego, California
  - Syrentis Clinical Research, Santa Ana, California
  - Colorado Medical Research Center, Denver, Colorado
  - The Savin Center, PC, New Haven, Connecticut
  - Altus Research, Lake Worth, Florida
  - The Miami Institute, Miami, Florida
  - Baumann Cosmetic and Research Institute, Miami, Florida
  - Miami Research Associates, South Miami, Florida
  - Clinical Research of West Florida, Inc., Tampa, Florida
  - DeNova Research, Chicago, Illinois
  - Laser and Skin Surgery Center of Indiana, Carmel, Indiana
  - South Bend Clinic, South Bend, Indiana
  - SkinCare Physicians, Chestnut Hill, Massachusetts
  - Zel Skin & Laser Specialist, LLC, Edina, Minnesota
  - Mercy Health Research, Washington, Missouri
  - Image Dermatology, Montclair, New Jersey
  - Sadick Research Group, New York, New York
  - Wake Research Associates, Raleigh, North Carolina
  - Oregon Medical Research Center, Portland, Oregon
  - Chaddsford Dermatology, Chadds Ford, Pennsylvania
  - Paddington Testing Co., Inc., Philadelphia, Pennsylvania
  - Society Hill Dermatology, Philadelphia, Pennsylvania
  - Tennessee Clinical Research Center, Nashville, Tennessee
  - DermResearch Inc., Austin, Texas
  - Modern Research Associates, PLLC, Dallas, Texas
  - Suzanne Bruce and Associates, P.A., The Center for Skin Research, Houston, Texas
  - Austin Institute Clinical Research, Pflugerville, Texas
  - Premier Clinical Research, Spokane, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- LIPO-202: Experimental arm
  LIPO-202
- Placebo: Placebo comparator
  Placebo
Period: Overall Study
Arm/Group | LIPO-202 | Placebo
Started | 398 | 395
Completed | 371 | 361
Not Completed | 27 | 34
Not completed — Adverse Event | 2 | 3
Not completed — Lost to Follow-up | 5 | 0
Not completed — Non-compliance | 4 | 4
Not completed — Protocol Violation | 6 | 10
Not completed — Sponsor Decision | 2 | 1
Not completed — Pregnancy | 1 | 0
Not completed — Withdrawal by Subject | 7 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LIPO-202 | Placebo | Total
Number analyzed (Participants) | 398 | 395 | 793
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (11.7) | 41 (12.2) | 40 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 327 | 334 | 661
  Male | 71 | 61 | 132
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 83 | 78 | 161
  Not Hispanic or Latino | 315 | 317 | 632
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 0 | 4
  Asian | 24 | 17 | 41
  Native Hawaiian or Other Pacific Islander | 1 | 3 | 4
  Black or African American | 36 | 37 | 73
  White | 316 | 325 | 641
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 17 | 13 | 30
Region of Enrollment [Number; unit: participants]
  United States | 398 | 395 | 793

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Who Achieved a Composite P-GAPS1/CPnS2 Response
Description: The composite P-GAPS1/CPnS2 response was defined as at least a 1 point (grade) improvement in P-GAPS and at least a 2 point (grade) improvement in CPnS from baseline after 8 weeks of treatment.
  Patient - Global Abdominal Perception Scale (P-GAPS) - a patient views and assesses the contour of their abdomen on a 5-point verbal scale ranging from "Flat" to "Big Bulge".
  Clinician Photonumeric Scale (CPnS) - a trained clinician rater examines the subject's abdomen and matches the subject's abdominal bulge/profile to the nearest gender-specific abdominal photo on the 6-point scale.
Time Frame: Baseline and End of Study (1 week post last treatment, 9 weeks after first treatment)
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | LIPO-202 | Placebo
Number analyzed (Participants) | 368 | 361
Participants | 37 | 48
Statistical Analysis 1: Comparison: LIPO-202 vs Placebo; Test type: Superiority; p = 0.397, Cochran-Mantel-Haenszel

2. Primary Outcome: Percent Change in the Patient Reported Global Abdominal Perception Score
Description: 1 equals much improved, 7 equals much worse. The higher the scores the worse the outcome.
Time Frame: 8 weeks post the start of treatment
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | LIPO-202 | Placebo
Number analyzed (Participants) | 398 | 395
percent change | 202 (51) | 175 (44)
Statistical Analysis 1: Comparison: LIPO-202 vs Placebo; Test type: Superiority; p = 0.379, Cochran-Mantel-Haenszel

3. Secondary Outcome: Percent Change in Waist Circumference
Time Frame: 8 weeks post the start of treatment
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | LIPO-202 | Placebo
Number analyzed (Participants) | 398 | 395
percent change | 24.1 (2.65) | 24.2 (2.66)

ADVERSE EVENTS:
Time Frame: The collection of adverse events from the first dose of study drug until the End-of-Study Visit (one week post last treatment) or at the Early Termination Visit.
Arm/Group | LIPO-202 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/398 | 0/395
Serious Adverse Events (participants affected / at risk) | 1/398 | 1/395
Other Adverse Events (participants affected / at risk) | 138/398 | 150/395
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LIPO-202 (N=398) | Placebo (N=395)
Ankle Fracture (Injury, poisoning and procedural complications) | 0 | 1
Cerebrovascular Accident (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LIPO-202 (N=398) | Placebo (N=395)
Injection Site Bruising (General disorders) | 107 | 110
Injection Site Haemorrhage (General disorders) | 13 | 13
Injection Site Pain (General disorders) | 10 | 15
Injection Site Erythema (General disorders) | 4 | 4
Upper Respiratory Tract Infection (Infections and infestations) | 4 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other